CLINICAL TRIAL: NCT01578616
Title: Association of Endothelial Function With Plaque Vulnerability Assessed by Optical Coherence Tomography in Patients With Acute Coronary Syndrome
Brief Title: Endothelial Dysfunction and Plaque Vulnerability
Status: Completed | Type: Observational
Sponsor: Yokohama City University Medical Center (Other)
Responsible Party: Principal Investigator, Kiyoshi Hibi, Associate Professor of Medicine, Yokohama City University Medical Center
Other Study IDs: RHI OCT study
Record Dates: First submitted 2012-04-11; First posted 2012-04-17 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Acute Coronary Syndrome
Keywords: Coronary artery disease; Endothelial function; Optical coherence tomography; Thin cap fibroatheroma
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 3 / non-CAD, ACS with or without TCFA: ACS patients with thin cap fibroatheroma. ACS patients without thin cap fibroatheroma. Age-, gender-, and rate of hypertension or diabetes mellitus-matched patients who have never been diagnosed or treated for CAD are also enrolled as non-CAD patients
- non-CAD, ACS without TCFA, ACS with TCFA: Acute coronary syndrome (ACS) patients with thin cap fibroatheroma. ACS patients without thin cap fibroatheroma. Age-, gender-, and rate of hypertension or diabetes mellitus-matched patients who have never been diagnosed or treated for CAD are also enrolled as non-CAD patients

SUMMARY:
Thinning of fibrous cap in atherosclerotic plaques is associated with plaque vulnerability. The high resolution of optical coherence tomography (OCT) provides an accurate measurement of fibrous cap thickness. Endothelial dysfunction is a key component of vulnerable plaque and digital reactive hyperemia-peripheral arterial tonometry (RH-PAT) is a non-invasive automatic and quantitative method to evaluate endothelial function. The investigators will investigate the association between endothelial function assessed by RH-PAT and plaque vulnerability determined by OCT-derived thin-cap fibroatheroma (TCFA).

DETAILED DESCRIPTION:
Consecutive patients with acute coronary syndrome (ACS) who undergo both OCT examination and RH-PAT examination are enrolled. OCT examination is performed to observe the culprit lesion before percutaneous coronary intervention, and endothelial function is evaluated using RH-PAT before discharge.

ELIGIBILITY:
Inclusion Criteria:

* patients with angiographically proven ACS (luminal stenosis of at least 50%) who undergo both OCT examination before coronary stent implantation and RH-PAT examination before discharge.

Exclusion Criteria:

* none

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Yokohama City University Medical Center
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kiyoshi Hibi, MD, PhD, Principal Investigator — Division of Cardiology, Yokohama City University Medical Center
Locations (1):
- Division of Cardiology, Yokohama City University Medical Center, Yokohama, Japan